CLINICAL TRIAL: NCT06682325
Title: Development of a Pharmaco-proteomic Platform to Evaluate Potential Drug Interactions and Their Clinical Impact in Liver Transplant Patients Undergoing Multidrug Treatment
Brief Title: Pharmaco-proteomic Platform to Evaluate Drug Interactions in Liver Transplant Patients
Status: Recruiting | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Universidad de Valparaiso (Other); Universidad Adolfo Ibañez (Unknown)
Responsible Party: Sponsor
Other Study IDs: 23I10401
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-07

CONDITIONS: Drug-drug Interaction; Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and serum samples from patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Other: Multi-drug interaction — The clinical impact associated with the use of multiple drugs in liver transplant patients during their stay in ICU will be evaluated.

SUMMARY:
The goal of this observational study is to enhance the ability to forecast kidney failure in liver transplant patients in the ICU under multidrug treatment by developing a computer platform that integrates mathematical models of drug interactions, proteomics, and clinical data. The main outcomes it aims to develop are:

1. Design the multidrug web computing platform with available information on drug pair interactions (DDIs).
2. Integrate the proteomic and clinical data of liver transplant patients into the IT platform.
3. Implement the multidrug web platform to predict the clinical evolution of liver transplant patients.

DETAILED DESCRIPTION:
The aim of this project is to enhance the ability to forecast kidney failure for liver transplant patients in the ICU by developing a computer platform that integrates mathematical models of drug interactions, proteomics, and clinical data. This integrated platform enables the prediction of the development of AKI in patients who have undergone OLT. Through the integration of mathematical models, the platform captures complex interactions between multiple drugs and proteomics data from patients, contributing to an improved predictive capacity for AKI outcomes.

By leveraging proteomic insights, personalized therapeutic interventions can be devised, promoting safer and more effective treatments. This research seeks to empower medical professionals with comprehensive information to navigate the complex landscape of drug interactions and personalized treatment strategies, ultimately contributing to improved patient outcomes and healthcare practices in the realm of liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant patients undergoing surgery at UC Christus Hospital

Exclusion Criteria:

* Patients on renal replacement therapy
* Patients for whom no clinical or pharmacological registry is available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant patients admitted to intensive care after surgery
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-05 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Develop a web platform that combines information on interactions between multiple drugs and proteomic and clinical profiles, to predict the clinical evolution in liver transplant patients hospitalized in the ICU | 18 to 24 months
  Periodic developmental assessments will be carried out (Analysis of drug interaction graphs, Design of the interaction web platform, Integration of omics and clinical data into the web platform)

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Barrera, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (3):
- Chile (3):
  - Universidad de Valparaíso, Valparaíso, Región de Valparaíso
  - Hospital ClínicoUC-Christus, Santiago, Santiago Metropolitan
  - Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: No